CLINICAL TRIAL: NCT06617962
Title: Evaluation of The Diagnostic Value of Two Cell-based Assays for MOG-IgG-associated Diseases: A Multicenter, Paired Design Observational Study
Brief Title: Evaluation of Two Cell-based Assays for Diagnosing MOG-IgG Associated Disorders
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chao Quan, Professor, Huashan Hospital
Other Study IDs: KY2024-1005
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Myelin Oligodendrocyte Glycoprotein (MOG)-Antibody Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study participants with high clinical suspicion of MOGAD: Based on the "Chinese Expert Consensus on the Diagnosis and Treatment of Myelin Oligodendrocyte Glycoprotein Immunoglobulin MOG-IgG Antibody Associated Diseases" and the "Diagnosis of myelin oligodendrocyte glycoprotein antibody-associated disease: International MOGAD Panel proposed criteria" in2023
  Interventions: Diagnostic Test: CBA method of live cells and fixed cells
- Control group: including 30 participants in the study of other inflammatory CNS diseases, 30 participants in the study of non-inflammatory CNS and 30 participants in the study of healthy people
  Interventions: Diagnostic Test: CBA method of live cells and fixed cells

INTERVENTIONS:
Diagnostic Test: CBA method of live cells and fixed cells — 1. Study participants with high clinical suspicion of MOGAD: 2mL serum samples were collected for detection. CBA method of live cells and fixed cells was used for all samples. Sensitivity, specificity, positive predictive value and negative predictive value of the two detection methods were calculated according to the detection results and combined with the 2023 MOGAD diagnostic criteria.
  2. Control group：2mL serum samples were collected for detection. CBA method of live cells and fixed cells was used for all samples.

SUMMARY:
Anti-myelin oligodendrocyte glycoprotein-IgG-associated disorders (MOGAD) is a rare inflammatory autoimmune disease. In addition, since the international MOGAD group proposed live-cell based assays for MOGAD diagnosis in 2023, there are still no real-world cohort validation studies on this methodology. This study intends to establish a large sample cohort with multi-center and paired design. MOG-IgG detection based on live cells and fixed cells was performed on the study participants with high suspicion of MOGAD and the negative control population, to obtain the diagnostic performance parameters and consistency evaluation of the two methodologies, evaluate their clinical diagnostic value, and explore the best individual assay cutoffs for MOG-IgG detection suitable for the diagnosis of MOGAD in China.

DETAILED DESCRIPTION:
Study design: A multicenter, observational study to compare the diagnosis performance of two cell-based assays in Chinese patients with idiopathic demyelinating disorders Participants: In this study, serum samples were collected from participants with high clinical suspicion of MOGAD (the number of valid positive cases was 150), and control samples were collected (including 30 participants in other inflammatory CNS disease studies, 30 participants in non-inflammatory CNS studies, and 30 participants in healthy people studies).

Aim: In this multicenter study, a cell-based assay (CBA) based on cell transfection was proposed to semi-quantitatively detect specific antibodies in human serum samples of study participants with highly suspected clinical manifestations of MOGAD and the control population. Each study participant used two CBA detection methods to detect MOG-IgG at the same time, namely live cell based and fixed cell based, to obtain diagnostic performance parameters and consistency evaluation (sensitivity, specificity, positive predictive value, negative predictive value) of the two methods, and combined with comprehensive clinical diagnosis to compare their clinical diagnostic value. To explore the individual assay cutoffs for the diagnosis of MOGAD in China.

Total enrollment: participants with high clinical suspicion of MOGAD (the number of valid positive cases was 150), and control samples were collected (including 30 participants in other inflammatory CNS disease studies, 30 participants in non-inflammatory CNS studies, and 30 participants in healthy people studies).

Time frame: August 1, 2024 to December 1, 2025.

Study protocol:

1. This study intends to include participants with a high likelihood of MOGAD, and to simultaneously match a negative control group including inflammatory CNS disease, non-inflammatory CNS disease, and healthy people. Serum samples of the above study participants were detected by CBA method of live cells and fixed cells. According to the comprehensive diagnosis results of clinical experts, the specificity, sensitivity, positive predictive value and negative predictive value of the two methods were compared, and the clinical consistency of the two methods was obtained.
2. According to the comprehensive clinical diagnosis results, the consistency of MOG-IgG positive and titer results between active CBA method and fixed CBA method was evaluated.
3. According to the comprehensive clinical diagnosis, the diagnostic value of MOGAD in different titers of the two methods was evaluated. To obtain the best individual assay cutoffs of MOGAD diagnosis in this study and improve the specificity of disease diagnosis.
4. The proportion of study participants with high suspicion of MOGAD who were diagnosed with MOGAD was counted, and the clinical characteristics of participants in this part of the study were analyzed to explore the correlation between MOG-IgG antibody titers and clinical characteristics, treatment regimen, clinical course, or disease activity.

Official Title Evaluation of the diagnostic value of two cell-based assays for MOG-IGG-associated diseases: a multicenter, paired design observational study Conditions MOG-IgG detection Intervention / Treatment Diagnostic Test: CBA method of live cells and fixed cells.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old, male and female.
* MOGAD is highly suspected.
* Other inflammatory CNS disease control groups include: According to the diagnostic criteria and consensus of various diseases, the diagnosis of multiple sclerosis, Autoimmune encephalitis (except NMDAR encephalitis), Guillain-Barre syndrome (GBS), Chronic Inflammatory Demyelinating polyradiculopathy (CIDP), Retinal Cerebrovascular disease (SUSAC), POEMS syndrome (POEMS), and neuropathy were confirmed. The monoclonal gammopathy of unknown significance (MGUS), Sarcoidosis and so on.
* The control group of non-inflammatory central nervous system diseases included: Migraine, CSVD, benign cranial hypertension, Glioma with definite diagnosis and no other autoimmune diseases.
* Healthy controls include healthy people who have no autoimmune diseases through physical examination and other means.
* Complete clinical data.
* Informed consent of the patient or his guardian has been obtained.

Exclusion Criteria:

* According to the Guidelines for Diagnosis and Treatment of Optic Neuromyelitis Spectrum Diseases (2021), patients with optic Neuromyelitis Spectrum diseases (NMOSD) with positive AQP4 were clearly diagnosed.
* According to the Expert Consensus on the Diagnosis and Treatment of Autoimmune encephalitis in China (2022), the diagnosis was confirmed as NMDAR encephalitis.
* Patients with positive anti-glial fibrillary acidic protein antibody (GFAP-IgG) in serum and/or cerebrospinal fluid.
* Lack of clinical data.
* Unqualified blood samples.
* The patient's informed consent was not obtained.
* Misdiagnosis in the research process went wrong in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individual medical units plan to collect serum samples from clinically suspected MOGAD study participants (150 valid positive cases will be the cutoff for sample collection) between September 2024 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance parameters and consistency evaluation | August 1, 2024 to December 1, 2025.
  Each study participant used two cell-based assays to detect MOG-IgG simultaneously, namely live cell based and fixed cell based, to obtain the diagnostic performance parameters and consistency evaluation (sensitivity, specificity, positive predictive value, negative predictive value) of the two methodologies.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Chao, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China